CLINICAL TRIAL: NCT04472442
Title: Intermittent Hypoxia Paired with High Intensity Training in Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Rehabilitation Hospital of Indiana (Other)
Responsible Party: Principal Investigator, George Hornby, Professor of Physcial Medicine & Rehabilitation, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IU2001598586
Record Dates: First submitted 2020-07-13; First posted 2020-07-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-05

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: 2-arm, randomized, crossover trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of both participant with actual vs sham treatment and blinding of primary outcome assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Intensity Training with Intermittent Hypoxia (Experimental): The primary goal will be provide acute intermittent hypoxia (9% PO2; 1 min on 1 min off) prior to stepping training while maintaining HR within 70-85% maximum predicted HR (if patients are deconditioned, PTs will gradually increase intensity to desired levels as tolerated). Sessions will be divided into ~10 minute increments (~25% of sessions) between speed-dependent treadmill training (described above for treadmill stepping), skill-dependent treadmill training, overground training, and stair climbing.
  Interventions: Procedure: Intermittent hypoxia
- High Intensity Training with Sham Hypoxia (Sham Comparator): The primary goal will be provide sham intermittent hypoxia (20% PO2) prior to performing continuous stepping while maintaining HR within 70-85% maximum predicted HR (if patients are deconditioned, PTs will gradually increase intensity to desired levels as tolerated). Sessions will be divided into ~10 minute increments (~25% of sessions) between speed-dependent treadmill training (described above for treadmill stepping), skill-dependent treadmill training, overground training, and stair climbing.
  Interventions: Procedure: Sham hypoxia

INTERVENTIONS:
Procedure: Intermittent hypoxia — Acute intermittent treatment (AIH) will be initiated using an oxygen generator (Model HYP-123, Hypoxico Inc, New York, NY, and participants will be seated comfortably and fitted with a non-rebreather mask. AIH (using 9% O2) will be provided in 60 s intervals and repeated 15 times with alternating 60 s intervals of normoxia (21% O2). Continuous pulse oximetry (Masimo 7, Irvine CA) will be monitored to ensure oxygen saturation of 82-85%. Signs and symptoms of distress with AIH exposure will be noted throughout, with HR and blood pressure taken every 3-5 minutes and documented.
  High-intensity training will then be performed (40 min of walking training up to 70-80% maximum heart rate within 1 hr).
  Arms: High Intensity Training with Intermittent Hypoxia
Procedure: Sham hypoxia — Sham acute intermittent treatment (sham AIH) will be initiated using an oxygen generator (Model HYP-123, Hypoxico Inc, New York, NY, and participants will be seated comfortably and fitted with a non-rebreather mask. Sham AIH (using 20% O2) will be provided in 60 s intervals and repeated 15 times with alternating 60 s intervals of normoxia (21% O2). Continuous pulse oximetry (Masimo 7, Irvine CA) will be monitored to ensure oxygen saturation of 82-85%. Signs and symptoms of distress with AIH exposure will be noted throughout, with HR and blood pressure taken every 3-5 minutes and documented.
  High-intensity training will then be performed (40 min of walking training up to 70-80% maximum heart rate within 1 hr).
  Arms: High Intensity Training with Sham Hypoxia

SUMMARY:
The central hypotheses are that HIT combined with AIH results in: 1) greater locomotor gains as compared to HIT alone; 2) improvements in gait quality and motor coordination during walking, and 3) changes in measures of community participation and integration.

DETAILED DESCRIPTION:
The central hypotheses are that HIT combined with AIH results in: 1) greater locomotor gains as compared to HIT alone; 2) improvements in gait quality and motor coordination during walking, and 3) changes in measures of community participation and integration. To test these hypotheses, the proposed crossover, assessor-blinded, randomized clinical trial (RCT) is designed to test the effects of safety, feasibility, and preliminary efficacy of HIT+AIH. In this phase I-II trial, patients >6 months post-BI with mobility deficits will be allocated to 5 weeks (15 sessions) of HIT+AIH or HIT alone. Blinded assessments will be performed prior to and following training paradigms to address 3 specific aims.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months post brain injury
* 18-85 years old
* ability to walk without physical assistance
* Self selected walking speed of 0.01-1.0 m/s

Exclusion Criteria:

* <18 years old
* >85 years old
* self selected walking speed of > 1.0 m/s
* < 3 months from botulinum toxin injection above the knee brace
* Currently receiving physical therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | Baseline 1, Post 1 after 6 weeks, Baseline 2, Post 2 after 6 weeks
  Gait speed is valid, reliable, and sensitive measures related to overall functional ability, and will be assessed by blinded rates. This measure will be performed by blinded assessors who do not participate in the training. Gait speed will be measured at self-selected speeds (SSS; instructions to "walk at normal comfortable pace") and fastest-possible speed (FS: "as fast as you safely can") using the Zeno Walkway (Protokinetics, Haverton, PA).
Change in Endurance | Baseline 1, Post 1 after 6 weeks, Baseline 2, Post 2 after 6 weeks
  Endurance is valid, reliable, and sensitive measures related to overall functional ability, and will be assessed by blinded rates. This measure will be performed by blinded assessors who do not participate in the training. Gait endurance will be tested using the 6MWT (m) with instructions similar to SSS to minimize fall risk.

SECONDARY OUTCOMES:
Metabolic capacity | Baseline 1, Post 1 after 6 weeks, Baseline 2, Post 2 after 6 weeks
  Peak metabolic capacity will be observed during graded exercise testing on a treadmill wtih peak oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hornby, PT,PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
IPD available per request

REFERENCES:
- [Derived] Hornby TG, Plawecki A, Lotter JK, Shoger LH, Voigtmann CJ, Inks E, Henderson CE. Acute Intermittent Hypoxia With High-Intensity Gait Training in Chronic Stroke: A Phase II Randomized Crossover Trial. Stroke. 2024 Jul;55(7):1748-1757. doi: 10.1161/STROKEAHA.124.047261. Epub 2024 Jun 11. PMID 38860389